CLINICAL TRIAL: NCT02281955
Title: De-intensification of Radiation and Chemotherapy for Low-Risk HPV-related Oropharyngeal Squamous Cell Carcinoma
Brief Title: De-intensification of Radiation and Chemotherapy for Low-Risk HPV-related Oropharyngeal SCC: Follow-up Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1413
Record Dates: First submitted 2014-10-03; First posted 2014-11-04 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms
Keywords: Human Papillomavirus; Oropharynx; Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma; Radiation Therapy; Chemotherapy; p16
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- De-escalated Radiation and Chemotherapy (Experimental): Patients will receive Intensity Modulated Radiotherapy Treatments (IMRT), 60 Gy at 2 Gy/fx. The acceptable weekly chemotherapy regimens are Cisplatin 30 to 40 mg/m2 (first choice), Cetuximab 250mg/m2 (second choice), Carboplatin AUC 1.5 and paclitaxel 45 mg/m2 (third choice), Carboplatin AUC 3 (fourth choice). Chemotherapy will be given intravenously weekly during IMRT, 6 total doses. Chemotherapy will not be given to patients with T0-2 N0-1 disease, ≤ 10 pack years smoking history. Decision for surgical evaluation will be based on the results of the PET/CT and clinical exam 10-16 weeks after CRT. Patients with a positive PET/CT scan will undergo surgical evaluation at the discretion of the surgeon. Patients with a negative PET/CT scan will be observed.
  Interventions: Radiation: Intensity Modulated Radiotherapy (IMRT); Drug: Cisplatin (or alternative); Procedure: Assessment for surgical evaluation

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy (IMRT) — All patients will receive Intensity Modulated Radiotherapy Treatments (IMRT). Dose painting IMRT will be used and all doses will be specified to the planning target volume (PTV). The high risk planning target volume (PTV-HR) and standard risk planning target volume (PTV-SR) will be treated to the following respective total doses: 60 Gy and 54 Gy. The dose per fraction to the PTV-HR and PTV-SR will be 2 Gy per day and 1.8 Gy per day respectively. The PTV-HR will include the gross tumor and the PTV-SR will include areas at risk for harboring subclinical microscopic disease.
Drug: Cisplatin (or alternative) — Cisplatin is the preferred mandated first choice chemotherapy, however alternative weekly regimens are permissible. Justification for not using cisplatin must be documented. Chemotherapy will be given intravenously weekly during IMRT. 6 total doses will be given. It is preferred that the doses be administered on days 1, 8, 15, 22, 29, and 36; however, this is not mandatory. Chemotherapy will not be given to patients with T0-2 N0-1 disease, ≤ 10 pack years smoking history.
Procedure: Assessment for surgical evaluation — Decisions for surgical evaluation will be based on the results of the PET/CT 10 to 16 weeks after CRT and clinical exam (including fiberoptic laryngoscopy) at that time. Other optional imaging studies may be performed. Patients with a positive PET/CT scan will undergo surgical evaluation at the discretion of the surgeon, with the goal being to remove any suspected residual tumor with a negative resection margin while maintaining organ preservation. This may include biopsies and/or oncological resections of the primary tumor and lymph node metastases. Patients with a negative PET/CT scan will be observed.

SUMMARY:
The purpose of this research study is to learn about the effectiveness of using lower-intensity radiation and chemotherapy to treat human papillomavirus (HPV) associated low-risk oropharyngeal and/or unknown primary squamous cell carcinomas of the head and neck. The cure rate for this type of cancer is estimated to be high, > 90%. The standard treatment for this cancer is 7 weeks of radiation with 3 high doses of cisplatin. Sometimes surgery is performed afterwards. This standard regimen causes a lot of side effects and long term complications. This study is evaluating whether a lower dose of radiation and chemotherapy may provide a similar cure rate as the longer, more intensive standard regimen. Patients in this study will receive 1 less week of radiation and a lower weekly dose of chemotherapy.

DETAILED DESCRIPTION:
The proposed study is a follow-up study to NCT01530997. In NCT01530997, patients with HPV positive and/or p16 positive low-risk oropharyngeal squamous cell carcinoma (OPSCC) received de-intensified chemoradiotherapy (CRT) followed by a limited surgical evaluation. The primary endpoint of NCT01530997 was the rate of pathological complete response (pCR) after CRT. Power computations were performed for N=40 and were based on the null hypothesis (H0) that the pCR for de-intensified chemoradiotherapy is at least 87%, the historical rate. The type 1 error for this calculation was 14.2%. 43 patients enrolled and 38 were evaluable for the primary endpoint. The observed pCR rate was 89% (34/38). Since the observed pCR rate was excellent in NCT01530997 and was in concordance with the expected rate, in the proposed study we will not mandate a post-CRT surgical evaluation. Instead a PET/CT 10 to 16 weeks post-CRT will be used to determine whether a surgical evaluation is needed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age (no upper age limit)
2. T0-3, N0 to N2c, M0 squamous cell carcinoma of the oropharynx
3. Biopsy proven squamous cell carcinoma that is HPV and/or p16 positive
4. ≤ 10 pack-years smoking history or ≤ 30 pack-years smoking history WITH ≥ 5 years abstinence from smoking
5. Radiologic confirmation of the absence of hematogenous metastasis within 12 weeks prior to treatment
6. ECOG Performance Status 0-1
7. CBC/differential obtained within 8 weeks prior to treatment, with adequate bone marrow function defined as follows: Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl.
8. Adequate renal and hepatic function within 4 weeks prior to registration, defined as follows: Serum creatinine < 2.0 mg/dl; Total bilirubin < 2 x the institutional ULN; AST or ALT < 3 x the institutional ULN.
9. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential
10. Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment.
11. Patients must be deemed able to comply with the treatment plan and follow-up schedule.
12. Patients must provide study specific informed consent prior to study entry

Exclusion Criteria:

1. Prior history of radiation therapy to the head and neck
2. Prior history of head and neck cancer.
3. Unresectable disease (e.g. immobile node on physical exam, nodal disease that radiographically involves the carotid arteries, nerves)
4. Currently taking Disease Modifying Rheumatoid Drugs (DMRDs)
5. Severe, active co-morbidity, defined as follows: Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; Transmural myocardial infarction within the last 6 months; Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (Note, however, coagulation parameters are not required for entry into this protocol); Pre-existing ≥ grade 2 neuropathy; Prior organ transplant; Systemic lupus; Psoriatic arthritis.
6. Known HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2024-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette Shen, MD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Health, High Point, North Carolina
  - Rex Healthcare, Raleigh, North Carolina

REFERENCES:
- [Derived] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652
- [Derived] Chera BS, Amdur RJ, Green R, Shen C, Gupta G, Tan X, Knowles M, Fried D, Hayes N, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Zevallos J, Blumberg J, Patel S, Kasibhatla M, Sheets N, Weissler M, Yarbrough W, Mendenhall W. Phase II Trial of De-Intensified Chemoradiotherapy for Human Papillomavirus-Associated Oropharyngeal Squamous Cell Carcinoma. J Clin Oncol. 2019 Oct 10;37(29):2661-2669. doi: 10.1200/JCO.19.01007. Epub 2019 Aug 14. PMID 31411949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolling institutions included University of North Carolina Hospitals (Chapel Hill, NC), University of Florida Hospitals (Gainesville, FL), Rex Hospital (Raleigh, NC), High Point Regional Health (High Point, NC), and Pardee Memorial Hospital (Hendersonville, NC).
Pre-assignment Details: 115 patients were accrued. One patient voluntarily withdrew prior to treatment. One patient died during treatment secondary to neutropenic sepsis.
Groups:
- De-escalated Radiation and Chemotherapy: All patients were treated with Intensity Modulated Radiotherapy (IMRT). The total dose to the high-risk regions was 60 Gy at 2 Gy per fraction, 30 fractions, 5 days a week, for 6 weeks. Fifty-four gray was delivered to anatomic regions at risk of subclinical disease as indicated. Unilateral radiotherapy was permitted in patients with well-lateralized tonsil primaries. Cisplatin 30 mg/m2 once per week was the mandated first-choice chemotherapy; however, alternative regimens once per week were permissible. Chemotherapy was given intravenously once per week, preferably on Mondays. Six weekly doses were given concurrently with radiation. Dose modifications were allowed as needed per the treating medical oncologist's discretion. If a patient could not tolerate cisplatin for more than 1 week, he or she was switched to an alternative regimen. Chemotherapy was not given to patients with T0-2 N0-1 disease (AJCC 7th edition).
Period: Overall Study
Arm/Group | De-escalated Radiation and Chemotherapy
Started | 114
Completed | 113
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 114
Age, Continuous [Mean (Full Range); unit: years] | 62 [37 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 104
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 114
Marital Status [Count of Participants; unit: Participants]
  Married | 90
  Unmarried | 23
  Unknown | 1
Tobacco Use [Count of Participants; unit: Participants]
  Never smoked | 54
  <= 10 pack-years | 38
  > 10 pack-years | 22
Primary Tumor Location [Count of Participants; unit: Participants]
  Tonsil | 52
  Base of tongue | 57
  Unknown primary | 5
T Stage [Count of Participants; unit: Participants] — From less to more severe:
  T0 = No evidence of primary tumor T1 = Tumor 2 cm or less in greatest dimension T2 = Tumor more than 2 cm but not more than 4 cm in greatest dimension T3 = Tumor more than 4 cm in greatest dimension or extension to lingual surface of epiglottis
  Participants
    T0 | 5
    T1 | 35
    T2 | 61
    T3 | 13
N Stage (AJCC 7th edition) [Count of Participants; unit: Participants] — From less to more severe:
  N0 = No regional lymph node metastasis N1 = Metastasis in a single ipsilateral lymph node, 3 cm or less in greatest dimension N2a = Metastasis in a single ipsilateral lymph node more than 3 cm but not more than 6 cm in greatest dimension N2b = Metastasis in multiple ipsilateral lymph nodes, none more than 6 cm in greatest dimension N2c = Metastasis in bilateral or contralateral lymph nodes, none more than 6 cm in greatest dimension
  Participants
    N0 | 18
    N1 | 16
    N2a | 5
    N2b | 57
    N2c | 18
N Stage (AJCC 8th edition) [Count of Participants; unit: Participants] — From less to more severe:
  N0 = No regional lymph node metastasis N1 = One or more ipsilateral lymph nodes, none larger than 6 cm N2 = Contralateral or bilateral lymph nodes, none larger than 6 cm
  Participants
    N0 | 18
    N1 | 78
    N2 | 18
HPV/p16 Status [Count of Participants; unit: Participants]
  HPV+/p16+ | 46
  HPV-/p16+ | 12
  HPV unknown/p16+ | 56

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Progression Free Survival After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: Progression Free Survival (PFS) was defined as the time from the beginning of treatment to cancer progression or death. The outcome measure will be reported as the proportion of patients with PFS at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 112
Participants | 99

2. Secondary Outcome: 2 Year Local Control (LC) Rate After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: The outcome measure will be reported as the proportion of patients with LC at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 111
Participants | 107

3. Secondary Outcome: 2 Year Regional Control (RC) Rate After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: The outcome measure will be reported as the proportion of patients with RC at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 112
Participants | 110

4. Secondary Outcome: 2 Year Local-regional Control (LRC) Rate After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: The outcome measure will be reported as the proportion of patients with LRC at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 111
Participants | 105

5. Secondary Outcome: 2 Year Distant Metastasis Free Survival (DMFS) Rate After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: The outcome measure will be reported as the proportion of patients with DMFS at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 112
Participants | 103

6. Secondary Outcome: 2 Year Overall Survival (OS) Rate After De-intensified Chemoradiotherapy (CRT) in Human Papilloma Virus (HPV)-Positive and/or p16 Positive Low-risk Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: The outcome measure will be reported as the proportion of patients who are still alive (overall survival) at 2 years post-treatment.
Time Frame: Two years after completion of CRT on last enrolled patient (Note: CRT duration is 6 weeks).
Population: Note that the count provided here represents actuarial data and thus does not match the all-cause mortality count in the Adverse Events module.
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 114
Participants | 106

ADVERSE EVENTS:
Time Frame: 2 years post-treatment
Description: Only Grade 3 and higher events were collected across all sites and are reported here.
Arm/Group | De-escalated Radiation and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 5/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 59/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De-escalated Radiation and Chemotherapy (N=114)
Anemia (Blood and lymphatic system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 26
Anxiety (Psychiatric disorders) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Depression (Psychiatric disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 25
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 21
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 28
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nausea (Gastrointestinal disorders) | 11
Neck edema (General disorders) | 1
Sepsis (Infections and infestations) | 2
Pain (General disorders) | 15
Oral pain (Gastrointestinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Syncope (Nervous system disorders) | 1
Respiratory, thoracic, and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT02281955/Prot_SAP_001.pdf